CLINICAL TRIAL: NCT02023307
Title: Use of the V-Loc Suture for Mid-Face Lifting in Short-flap Rhytidectomy
Brief Title: Use of V-Loc Suture for Mid-face Lifting in Short-flap Rhytidectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinic Closed
Sponsor: Lifestyle Lift (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20131586
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Use of the Vloc Suture; Elevation of the Mid-face

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rhytidectomy with Covidien (Experimental): 25 patients receiving a mid-face lift in short-flap rhytidectomy
  Interventions: Device: V-Loc Suture

INTERVENTIONS:
Device: V-Loc Suture
  Other Names: Covidien

SUMMARY:
This study will evaluate and measure the Vloc suture's ability to elevate the mid-face when using a short flap, short incision technique in during a traditional face-lift. The objective of this study is to assess the suture's potential in elevating the mid-face when a traditional Lifestyle facelift is performed. We hypothesize that the Vloc suture will elevate the mid-face more effectively when using a short flap, short incision technique on a traditional facelift.

DETAILED DESCRIPTION:
A total of 25 patients who are already receiving a traditional Lifestyle Lift will be asked to participate. Once the consent form has been signed by the patient, the facelift will be performed as scheduled and the Vloc suture will be added to the mid-face area. Each patient will be added to a database and their progress will be tracked with photos taken before, at 6 weeks, and at 6 months following the procedure. All data stored will be locked into a hard drive that can only be accessed by the research staff and the doctor. The text data will be used by research staff for reports and articles.

* you must already have purchased and scheduled a facelift procedure with Lifestyle Lift to participate in this trial. The addition of only the V-loc suture is at no cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to receive a Lifestyle Lift will be asked to participate. The first 25 patients who have consented will be included into the study.

Exclusion Criteria:

* Any patient who is not able to receive a facelift for whatever reason, or who do not want a facelift will not be apart of this study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Elevation of the mid-face | Initial- 6 weeks

SECONDARY OUTCOMES:
No Retention of Mid-face | initial-6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Lifestyle Lift, Albuquerque, New Mexico, United States